CLINICAL TRIAL: NCT01234090
Title: Living With Aphasia: An International Study
Status: Terminated | Type: Observational
Why Stopped: Funding stopped
Sponsor: NYU Langone Health (Other)
Collaborators: The Solomon Foundation (Other); The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: 10-01628
Record Dates: First submitted 2010-10-15; First posted 2010-11-04 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Aphasia
Keywords: Aphasia; Quality of Life
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Persons with Aphasia

SUMMARY:
This prospective cohort study hypothesizes that an analysis of parallel qualitative and quantitative data is necessary to examine the full experience of living with aphasia. It is also hypothesized that there are specific factors that act as barriers or facilitators to successfully living with aphasia. A unique aspect of the project is the use of the Assessment for Living with Aphasia (ALA), a new aphasia friendly measure based on the World Health Organization International Classification of Functioning, Disability and Health (WHO ICF). Each session will assess written and spoken language, functional communication, mobility, Activities of Daily Living (ADL) function, burden of stroke, quality of life, and depression.

DETAILED DESCRIPTION:
Synopsis: This three year longitudinal study, based on a gerontological model, was the product of an Aphasia Think-Tank established in Toronto in 2007. The original concept and design, developed at Queensland Hospital in Australia, has been recently funded by the Australian National Health and Medical Research Council.

Rationale: Aphasia, which occurs in 30% of ischemic first strokes, is known to have a negative impact on quality of life, increase the incidence of post-stroke depression, be associated with a loss of self identity, and have a widespread effect on partners, children, siblings, and friends. Research conducted in Australia and the United Kingdom (UK) provides evidence that many persons living successfully with aphasia do not attribute their successes to speech-language pathology and rehabilitation services. Inappropriate, irrelevant, inaccessible, or non-existent required services have been cited. It has also been reported that current speech-language pathology service providers lack an overall understanding of the long term goals of aphasia rehabilitation and how these objectives may be achieved.

Hypothesis: It is hypothesized that an analysis of parallel qualitative and quantitative data is necessary to examine the full experience of living with aphasia; it is also hypothesized that there are specific factors that act as barriers or facilitators to successfully living with aphasia.

Methodology: The primary study site of this international research is the Community Disability Centre of the School of Health and Rehabilitation Medicine, University of Queensland. The Department of Rehabilitation Medicine, New York University (NYU) School of Medicine will collaborate by following, to the extent possible, the same protocols as the Australian team with respect to subject selection criteria, measures used, and test time-points. This is a prospective cohort study which uses parallel qualitative and quantitative (mixed) methods in a unique way to quantify the extent of and statistically model the relationship of the determinants to self-rated "successfully living with aphasia". Furthermore, it will permit an understanding of the underlying reasons (the why and how) behind the relationships. A unique aspect of the project is the use of the Assessment for Living with Aphasia (ALA), a new, aphasia friendly measure based on the World Health Organization International Classification of Functioning, Disability and Health (WHO ICF). It is a specialized tool using a self-rating scale and is focused on specific themes that have emerged from previous research. 204 subjects will be recruited who consent to being examined at 3, 6, and 12 months post-stroke. Considering an attrition rate of 25%, it is estimated that 153 subjects will provide the study data. Each session will be videotaped and consist of the administration of a demographic questionnaire, the Assessment for Living with Aphasia (ALA), the Western Aphasia Battery-Revised (a standardized measure which investigates language understanding and expression), a social-convoy model, the Barthel Index, the Wepman Self-Correction Scale, and the Aphasic Depression Rating Scale.

Anticipated Results: The outcomes of this project will lead to better services for people with aphasia via a fully articulated model of the predictive factors of success following aphasia. Not only will a statistical model be generated but the meaning of the factors and the relationships between them will be explained through the qualitative studies. For example, if decreasing social network size and satisfaction is a significant predictor variable of successfully living with aphasia, then rehabilitation services must target the loss of social networks in the first year through a variety of available but infrequently used interventions (e.g. communication partner training. The qualitative data will describe how social networks have changed (e.g. less contact with friends or formal groups) and why (e.g. communication or mobility issues) so that appropriate interventions are targeted to the correct group. This research will lead to substantial changes across the continuum of all aphasia rehabilitation services throughout the United States. Specifically, it will improve meaningful outcomes for persons with aphasia in terms of how to live successfully with aphasia. Results will also streamline aphasia services so that they meet the needs of this seriously disabled population who often cannot speak for themselves and rely on costly services for many years after their stroke. This international project will lead the way in changing speech pathology practices to meet the needs of people with aphasia around the world.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older, willingness to be videotaped, first incidence of aphasia secondary to stroke with stroke onset ≤2.5
* months pre-stroke or 3.5 months post-stroke with no significant complicating concomitant conditions (e.g. dementia, schizophrenia),
* premorbid fluency/literacy in English, and no history of psychiatric disorder, and sufficient communication ability (including adequate hearing and vision) in English to participate in an interview as determined by a qualified speech pathologist based on administration of the Western Aphasia Battery - Revised and clinical observation.
* participants will be enrolled in the study at 3 months post onset (+/- 2 weeks) wherever they are living, and presence of aphasia will be confirmed at the beginning of the first interview using the Aphasia Quotient cut offs of the Western Aphasia Battery.
* participants with severe global aphasia will only be excluded after the interview if meaningful responses cannot be obtained using all available communication support tools. Hence, participants with a range of aphasia severity will be included.

Exclusion Criteria:

* unwillingness to be videotaped
* onset of stroke <2.5 months post and >3.5 months post
* moderate or severe dementia
* symptoms of another preexisting neurological condition other than or in addition to aphasia due to stroke, or drug abuse
* neurological surgical treatment not including a surgical treatment specifically for treatment of stroke, absence of aphasia.
* no subjects will have a hearing loss unexpected for his/her chronological age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient/outpatient hospital population
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The Assessment for Living with Aphasia | 9 months
  A new, aphasia friendly measure based on the World Health Organization International Classification of Functioning, Disability, and Health. It is a specialized tool using a self-rating scale and is focused on specific themes that have emerged from previous research.

SECONDARY OUTCOMES:
Western Aphasia Battery - Revised | 9 months
  This measure is designed to assess clinical aspects of language functions in aphasic patients and to provide the data needed to establish a prognosis for therapy.
Successfully Living with Aphasia Rating Scale | 9 months
  This scale is a quantitative self-rating of how successfully a person is living with aphasia.
Burden of Stroke Scale | 9 months
  The Burden of Stroke Scale is a health-status assessment instrument designed to measure patient-reported difficulty in multiple domains of functioning, psychological distress associated with specific functional limitations, and general well-being in stroke survivors.
Aphasia Depression Rating Scale | 9 months
  The Aphasic Depression Rating Scale (ADRS) was developed to detect and measure depression in aphasic patients during the subacute stage of stroke.
The Wepman Self-Correction Scale | 9 months
  This scale, based on a continuum, measures disturbances in the ability of the person with aphasia to self-correct speech and language errors.
The Barthel Index | 9 months
  This measure is a simple index of independence to score the ability of a patient with a neuromuscular or musculoskeletal disorder to care for himself.
The Functional Communication Profile | 9 months
  This rating scale is for persons with aphasia which considers 45 everyday communication behaviors. Ratings of each behavior are made on a 9-point scale, based on observations of the patient during an informal conversation.

CONTACTS AND LOCATIONS:
Overall Officials: Martha T Sarno, MA,Dhonorary, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States